CLINICAL TRIAL: NCT02173938
Title: Novel Psychosocial Influences on Successful Tobacco Cessation Among Treatment Seekers
Brief Title: Novel Psychosocial Influences on Smoking Cessation
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Michael B. Steinberg, MD, MPH, FACP, Associate Professor of Medicine, Rutgers, The State University of New Jersey
Other Study IDs: CINJ#131217
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Smoking
Keywords: Smokers; outpatient; Tobacco Dependence Treatment Program
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment seekers
  Interventions: Other: Tobacco Dependence Treatment

INTERVENTIONS:
Other: Tobacco Dependence Treatment — face to face, outpatient tobacco dependence treatment based on the Public Health Service guidelines for treating tobacco use and dependence

SUMMARY:
Our overall research goal is to determine how these novel psychosocial factors impact cessation. This pilot study will answer how dual use of other tobacco products, direct to consumer marketing, and the new phenomenon of butting-out and relighting influences cessation, and how understanding impulsivity and task persistence could lead to new and improved behavioral interventions for tobacco dependence. Answers to these pilot questions will lead to the publication of several manuscripts and provide important feasibility data to design large, well-powered clinical trials, population-level epidemiological studies, and contribute to furthering the field of tobacco treatment.

ELIGIBILITY:
Inclusion Criteria:

* smokers 18 years of age or older

Exclusion Criteria:

* non-English speaking participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult smokers 18 years and older seeking treatment for quitting smoking
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2012-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who have quit smoking | 6 months post quit date

CONTACTS AND LOCATIONS:
Locations (1):
- Tobacco Dependence Program, Rutgers University, New Brunswick, New Jersey, United States